CLINICAL TRIAL: NCT05043272
Title: Safety and Immune Response of COVID-19 Vaccination in Overweight People With Excessive BMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-76
Record Dates: First submitted 2021-09-10; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Overweight
Keywords: COVID-19
MeSH Terms: conditions — COVID-19; Overweight | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Overweight population with basic diseases: Basic diseases include diabetes, hypertension.
  Interventions: Biological: SARS-COV-2 VACCINE
- Overweight population with chronic liver diseases: Chronic liver diseases include chronic hepatitis ,liver cirrhosis, primary hepatocellular carcinoma.
  Interventions: Biological: SARS-COV-2 VACCINE
- Healthy population: Control group
  Interventions: Biological: SARS-COV-2 VACCINE

INTERVENTIONS:
Biological: SARS-COV-2 VACCINE — The antibody titer and adverse reactions were observed.

SUMMARY:
On 11 February 2020, the International Committee for the Classification of Viruses named the disease caused by SAＲS-CoV-2 infection in humans as the new coronavirus pneumonia (coronavirus disease 2019, COVID-19). Due to the changes of immune function and cardiopulmonary function in overweight people, the infection and severity of these patients are higher than that of the general population during the epidemic period. More attention should be paid to personal protection and disease prevention. Vaccination with COVID-19 vaccine can effectively prevent COVID-19 infection, delay or prevent patients from developing into critical illness and reducing mortality. In order to evaluate the safety and efficacy of COVID-19 vaccine for overweight people, and to guide COVID-19 vaccination more scientifically, rationally and effectively, this study was carried out.

DETAILED DESCRIPTION:
Due to the changes of immune function and cardiopulmonary function in overweight people, the infection and severity of these patients are higher than that of the general population during the epidemic period. More attention should be paid to personal protection and disease prevention. Vaccination of COVID-19 can effectively prevent COVID-19 virus infection and delay or prevent patients from developing into critical illness and reduce mortality. The safety and effectiveness of COVID-19 vaccine in this population were evaluated in order to play a scientific and theoretical supporting role in guiding COVID-19 vaccination more scientifically, reasonably and effectively. The samples of this study were collected and tested in the second affiliated Hospital of Chongqing Medical University. Patients with contraindications for vaccination will be excluded. The detected indexes included blood routine test, liver function, COVID-19 antibody titer, antibody duration and other indexes of healthy people (control group) and overweight people after vaccination ( 1, 3, 6 months after vaccination). The adverse reactions related to the vaccine were recorded.

ELIGIBILITY:
Inclusion Criteria:

- 1.Healthy group were as follows: no history of hepatitis, no history of liver cirrhosis, no history of liver cancer and receiving the whole-course COVID-19 vaccination.

2. Overweight people are defined as having a BMI of more than 24 and receiving the whole-course COVID-19 vaccination.

Exclusion Criteria:

* Patients previously diagnosed or with a history of contact with confirmed cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Overweight population with liver diseases or other basic diseases vaccinated with SARS-Cov-2 vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events after injection. | 1 month after vaccination
  The vaccine-related adverse reactions (such as fever, dizziness, fatigue, myalgia, etc.) were recorded and its safety was evaluated.
Number of participants with adverse events after injection. | 3 months after vaccination
  The vaccine-related adverse reactions (such as fever, dizziness, fatigue, myalgia, etc.) were recorded and its safety was evaluated.
Number of participants with adverse events after injection. | 6 months after vaccination
  The vaccine-related adverse reactions (such as fever, dizziness, fatigue, myalgia, etc.) were recorded and its safety was evaluated.

SECONDARY OUTCOMES:
Titer and duration of COVID-19 antibody production after vaccination | 1 month after vaccination
  The titer and duration of COVID-19 antibody were produced at 1 month
Titer and duration of COVID-19 antibody production after vaccination | 3 months after vaccination
  The titer and duration of COVID-19 antibody were produced at 3 months
Titer and duration of COVID-19 antibody production after vaccination | 6 months after vaccination
  The titer and duration of COVID-19 antibody were produced at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ren, PH D, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- China, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Zhang C, Shi L, Wang FS. Liver injury in COVID-19: management and challenges. Lancet Gastroenterol Hepatol. 2020 May;5(5):428-430. doi: 10.1016/S2468-1253(20)30057-1. Epub 2020 Mar 4. No abstract available. PMID 32145190
- [Background] Grohskopf LA, Alyanak E, Broder KR, Walter EB, Fry AM, Jernigan DB. Prevention and Control of Seasonal Influenza with Vaccines: Recommendations of the Advisory Committee on Immunization Practices - United States, 2019-20 Influenza Season. MMWR Recomm Rep. 2019 Aug 23;68(3):1-21. doi: 10.15585/mmwr.rr6803a1. PMID 31441906
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Xu X, Sun J, Nie S, Li H, Kong Y, Liang M, Hou J, Huang X, Li D, Ma T, Peng J, Gao S, Shao Y, Zhu H, Lau JY, Wang G, Xie C, Jiang L, Huang A, Yang Z, Zhang K, Hou FF. Seroprevalence of immunoglobulin M and G antibodies against SARS-CoV-2 in China. Nat Med. 2020 Aug;26(8):1193-1195. doi: 10.1038/s41591-020-0949-6. Epub 2020 Jun 5. PMID 32504052
- [Result] Shi Q, Hu Y, Peng B, Tang XJ, Wang W, Su K, Luo C, Wu B, Zhang F, Zhang Y, Anderson B, Zhong XN, Qiu JF, Yang CY, Huang AL. Effective control of SARS-CoV-2 transmission in Wanzhou, China. Nat Med. 2021 Jan;27(1):86-93. doi: 10.1038/s41591-020-01178-5. Epub 2020 Nov 30. PMID 33257893
- [Result] Long QX, Tang XJ, Shi QL, Li Q, Deng HJ, Yuan J, Hu JL, Xu W, Zhang Y, Lv FJ, Su K, Zhang F, Gong J, Wu B, Liu XM, Li JJ, Qiu JF, Chen J, Huang AL. Clinical and immunological assessment of asymptomatic SARS-CoV-2 infections. Nat Med. 2020 Aug;26(8):1200-1204. doi: 10.1038/s41591-020-0965-6. Epub 2020 Jun 18. PMID 32555424
- [Result] Long QX, Liu BZ, Deng HJ, Wu GC, Deng K, Chen YK, Liao P, Qiu JF, Lin Y, Cai XF, Wang DQ, Hu Y, Ren JH, Tang N, Xu YY, Yu LH, Mo Z, Gong F, Zhang XL, Tian WG, Hu L, Zhang XX, Xiang JL, Du HX, Liu HW, Lang CH, Luo XH, Wu SB, Cui XP, Zhou Z, Zhu MM, Wang J, Xue CJ, Li XF, Wang L, Li ZJ, Wang K, Niu CC, Yang QJ, Tang XJ, Zhang Y, Liu XM, Li JJ, Zhang DC, Zhang F, Liu P, Yuan J, Li Q, Hu JL, Chen J, Huang AL. Antibody responses to SARS-CoV-2 in patients with COVID-19. Nat Med. 2020 Jun;26(6):845-848. doi: 10.1038/s41591-020-0897-1. Epub 2020 Apr 29. PMID 32350462
- See also: World Health Organization (WHO) Influenza (Seasonal) 2018 Available from — http://who.int/en/news-room/fact-sheets/detail/influenza-(seasonal)